CLINICAL TRIAL: NCT01324050
Title: Internet-delivered Psychodynamic Therapy for Depression: a Randomized Controlled Trial
Brief Title: Internet-delivered Psychodynamic Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Gerhard Andersson/Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-DEP2011-PDT
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internet-based Psychodynamic Therapy (Experimental)
  Interventions: Behavioral: Internet-delivered psychodynamic therapy for depression
- Internet-delivered therapist support (Active Comparator)
  Interventions: Behavioral: Internet-delivered therapist support

INTERVENTIONS:
Behavioral: Internet-delivered psychodynamic therapy for depression — This intervention contains 9 text-based self-help modules. These modules contain material inspired by psychoanalytic theory about identifying reoccurring patterns in life among other things. In addition to the self-help modules, 10-15 minutes of therapist contact is given every week. In total, the intervention will last for 10 weeks.
  Arms: Internet-based Psychodynamic Therapy
Behavioral: Internet-delivered therapist support — This intervention contains 1 text-based self-help module, which is mainly based on information on depression. In addition to this text, the participants in this group gets 10-15 minutes of therapist contact every week. In the conversation with the therapist, the participant informs the therapist about the activities during the week. This intervention is considered to be a form of support. In total, the intervention will last for 10 weeks.
  Arms: Internet-delivered therapist support

SUMMARY:
The overall aim of this study is to develop and test a psychodynamic Internet-delivered psychological treatment for patients with mild to moderate major depression and compare its efficacy to an active control group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder
* 15 or more on MADRS-S

Exclusion Criteria:

* Severe depression (more than 35 on MADRS-S or based on interview)
* Severe psychiatric condition (e.g. psychosis or bipolar disorder)
* Suicidal (measured in diagnostic interview)
* Changed medication during the last three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | Two weeks before the treatment starts
Beck Depression Inventory (BDI) | At treatment start (0 weeks)
Beck Depression Inventory (BDI) | At treatment termination (10 weeks)

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Two weeks before the treatment starts
Beck Anxiety Inventory (BAI) | At treatment termination (10 weeks)
Montgomery Åsberg Depression Rating Scale Self-report (MADRS-S) | Two weeks before treatment starts
Montgomery Åsberg Depression Rating Scale Self-report (MADRS-S) | At treatment termination (10 weeks)
Quality of Life Inventory (QOLI) | Two weeks before treatment starts
Quality of Life Inventory (QOLI) | At treatment termination (10 weeks)
Patient Health Questionnaire 9 (PHQ-9) | Two weeks before treatment starts
Patient Health Questionnaire 9 (PHQ-9) | At treatment termination (10 weeks)
Generalised Anxiety Disorder Assessment 7 (GAD-7) | Two weeks before treatment starts
Generalised Anxiety Disorder Assessment 7 (GAD-7) | At treatment termination (10 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Department of Behavioral Sciences and Learning, Linköping University
Locations (2):
- Sweden (2):
  - Linköping University, Department of Behavioral Sciences and Learning, Linköping
  - Linköping University, Linköping

REFERENCES:
- [Derived] Johansson R, Nyblom A, Carlbring P, Cuijpers P, Andersson G. Choosing between Internet-based psychodynamic versus cognitive behavioral therapy for depression: a pilot preference study. BMC Psychiatry. 2013 Oct 18;13:268. doi: 10.1186/1471-244X-13-268. PMID 24139066
- [Derived] Johansson R, Ekbladh S, Hebert A, Lindstrom M, Moller S, Petitt E, Poysti S, Larsson MH, Rousseau A, Carlbring P, Cuijpers P, Andersson G. Psychodynamic guided self-help for adult depression through the internet: a randomised controlled trial. PLoS One. 2012;7(5):e38021. doi: 10.1371/journal.pone.0038021. Epub 2012 May 29. PMID 22741027